CLINICAL TRIAL: NCT02726061
Title: Internet Based Psychological Support
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Jay C. Buckey Jr., Professor of Medicine, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00028777
Record Dates: First submitted 2016-02-29; First posted 2016-04-01 (Estimated); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Depression; Stress; Conflict Resolution
MeSH Terms: conditions — Depression; Negotiating

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Internet Based psychological support (Experimental): The internet-based psychological support intervention (PATH) is an internet based Problem Solving Therapy, stress management training and conflict management training program.
  Interventions: Behavioral: Internet-based psychological support

INTERVENTIONS:
Behavioral: Internet-based psychological support — A behavioral therapy called Problem Solving Therapy, conflict management training, and stress management training will be administered via an interactive multimedia program (PATH) to participants referred from their Employee Assistance Program and the general public for the management of depression, stress, and conflict.
  Other Names: PATH

SUMMARY:
The investigators have developed interactive, multimedia-intensive, computer-based treatment programs that include depression (Problem-Solving Therapy), stress management, and conflict management. Together the three modules are called PATH.

The problem-solving module is based on an evidence-based psychotherapy called Problem-Solving Therapy in which depressed patients identify problems in their lives and work through a structured format for solving these problems. We have subjected the problem-solving module to Phase 1-3 feasibility, acceptability and efficacy trials which have been positive and without adverse events.

The conflict program uses a cognitive-behavioral-therapy-based approach. The program includes a conflict briefing, an interactive conflict simulation, a conflict assessment tool, an interactive training exercise in interest-based negotiation, and a cognitive restructuring exercise.

The stress program also uses a cognitive behavioral therapy (CBT) approach. In the program, the mentor introduces the "stress pyramid", which demonstrates how stress triggers can lead to different feelings, actions and thoughts, which are analogs to the CBT realms of dysfunctional emotions, maladaptive behaviors, and faulty cognitive processes. The stress management content is delivered over 6 sessions, with each session including exercises in the 3 domains of thoughts, feelings, and actions. The program includes briefings, cognitive restructuring exercises, interactive scenarios, and self-assessments. This program has been evaluated with law and business students and was shown effective in reducing stress levels.

The purpose of the current study is to make the problem-solving, stress, and the conflict modules available through the internet for any adult 18 or older in order to assess their feasibility, acceptability and effectiveness under naturalistic conditions.

DETAILED DESCRIPTION:
Objective: To assess the feasibility, acceptability and effectiveness of PATH under naturalistic conditions.

Hypotheses:

H1: Greater than 50% of users referred to the problem-solving module will complete at least 4 treatment sessions.

H2: Users will report that problem-solving module is acceptable as a stand-alone treatment for depression.

H3: On average, user's self-reported depression severity scores on the PHQ-9 will decrease over time.

H4: More workers and family members will access the program directly than through referral from a clinician.

H5: Users will find the stress and conflict content acceptable and helpful in learning better stress and conflict management skills.

H6: On average, user self-reported stress severity scores on the PSS will decrease over time.

Procedures:

Consecutive employees and faculty members receiving evaluations in the EAP programs of Dartmouth-Hitchcock Medical Center (DHMC) and Dartmouth College and identified as being depressed or having issues with conflict or stress and as potentially able to benefit from using PATH will be referred to the program.

The programs are also available to any adult on their own or through their organization at:

Path.Dartmouth.edu

When the user signs up, they create a username and password and select they do not have a token and then are presented with an electronic consent. When they click accept (providing consent), they are given access to the programs.

Materials: PATH programs available on the internet.

Data Collection:

All study data will be automatically collected by the suite of programs (problem-solving, stress management, conflict management). Evaluation data (i.e., PHQ-9 scores and acceptability of the program) will be collected at each session. Information entered into the program as part of using PATH (e.g., the types of problems worked on, success with solving the problems, satisfaction with effort, compliance with homework, obstacles encountered) will also be automatically stored. Stress and conflict management programs collect the user input, the paths they take, and evaluation data. Users will create a login that will enable their use of the program.

The web-based programs are hosted at Dartmouth College. The web-app has passed an Acunetix security scan, run by Dartmouth Central Computing. It has been set up as a DISC level 3 security server. This has been evaluated by the Research Privacy and Security Officer at Dartmouth College and has been approved for use. Only gender will be collected. No identifying information (e.g., name, address, dob, SS#) will be collected. All entered data will be stored according to the assigned ID. To monitor for potentially nefarious hackers, IP addresses connecting to our servers will be collected and geo-located to ensure the router or internet service provider they are connecting from corresponds to those expected based on our research locations.

We do not propose to screen the participants for the study. Participants will be referred to the programs by their EAP counselor at Dartmouth-Hitchcock Medical Center, their FEAP counselor at Dartmouth College, their provider at DHMC, or by advertisement through Live Well Work Well or Dartmouth College EAP. Participants may also be referred through an outside organization or use the program on their own. As an effectiveness study, we are interested in making the programs available without exclusions to the general population. There are no eligibility criteria based on severity level of depression or suicidal ideation. There are no exclusion criteria for participation in the study. Suicidality is not a reason for not being enrolled in the study.

The program is being made available to Geisel Medical Students, as well as Dartmouth College and Dartmouth Hitchcock Employees through the Employee Assistance Program (EAP) at Dartmouth-Hitchcock Medical Center (DHMC), the Faculty and Employee Assistance Program (FEAP) at Dartmouth College and their D-H primary care physicians in order to assess their feasibility, acceptability and effectiveness under naturalistic conditions. Additionally, to test whether workers and their families are likely to access on-line treatment if they can access the treatment directly, we will make it possible for participants to connect to the programs directly, without referral from a clinician. We will be additionally testing these programs through making them freely available on the internet as well as through organizations that express interest in using them with their employees, members, etc. who are 18 or older.

Participants from outside of Dartmouth populations will be self-referred or referred to the program by people in their organization. We will not direct how the organizations will implement use of the programs but will collect information from the organizations about their implementation strategies. We may share usage data with the organizations but will not provide information for specific individuals.

For these populations, we will be analyzing usage data (i.e. completion of modules, return visits to modules), data collected by the program (i.e. progress through the modules), acceptability (i.e. from the questionnaires embedded in the programs such as the depression program), effectiveness (i.e. for those programs that include repeated assessments), and implementation strategies from different organizations that partner with us to use the program (i.e. reminder systems, adjunctive use with therapist, use in group settings).

ELIGIBILITY:
Inclusion Criteria:

* Adult employees (age 18 and older) and faculty attending the EAP programs of DHMC and Dartmouth College complaining of depression.
* Any Adult (age 18 or older)

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2016-02 (Actual); Primary Completion 2031-02 (Estimated); Study Completion 2031-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants referred to the PATH program that log on to the program. | Five years
  Does the participant log on to the program? yes/no

SECONDARY OUTCOMES:
Participant reports of the acceptability of the PATH program | Five years.
  Acceptability questionnaire

OTHER OUTCOMES:
Participant self-reported depression severity scores on the PHQ-9. | Five years
  Change in self-reported PHQ-9 score over time.
Participant self-reported stress severity scores on the PSS | Five years
  Change in self-reported PSS score over time

CONTACTS AND LOCATIONS:
Overall Officials: Jay C Buckey, M.D., Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sandoval LR, Buckey JC, Ainslie R, Tombari M, Stone W, Hegel MT. Randomized Controlled Trial of a Computerized Interactive Media-Based Problem Solving Treatment for Depression. Behav Ther. 2017 May;48(3):413-425. doi: 10.1016/j.beth.2016.04.001. Epub 2016 May 3. PMID 28390503
- [Background] Berman MI, Buckey JC Jr, Hull JG, Linardatos E, Song SL, McLellan RK, Hegel MT. Feasibility study of an interactive multimedia electronic problem solving treatment program for depression: a preliminary uncontrolled trial. Behav Ther. 2014 May;45(3):358-75. doi: 10.1016/j.beth.2014.02.001. Epub 2014 Feb 7. PMID 24680231
- [Background] Rose RD, Buckey JC Jr, Zbozinek TD, Motivala SJ, Glenn DE, Cartreine JA, Craske MG. A randomized controlled trial of a self-guided, multimedia, stress management and resilience training program. Behav Res Ther. 2013 Feb;51(2):106-12. doi: 10.1016/j.brat.2012.11.003. Epub 2012 Nov 21. PMID 23262118
- [Background] Anderson AP, Fellows AM, Binsted KA, Hegel MT, Buckey JC. Autonomous, Computer-Based Behavioral Health Countermeasure Evaluation at HI-SEAS Mars Analog. Aerosp Med Hum Perform. 2016;87(11):912-920. doi: 10.3357/AMHP.4676.2016. PMID 27779949
- [Derived] Detweiler Guarino I, Cowan DR, Fellows AM, Buckey JC. Use of a Self-guided Computerized Cognitive Behavioral Tool During COVID-19: Evaluation Study. JMIR Form Res. 2021 May 31;5(5):e26989. doi: 10.2196/26989. PMID 33973856
- See also: Internet-based psychological support (PATH) website — http://path.dartmouth.edu